CLINICAL TRIAL: NCT02286518
Title: A Single-center, Single- and Multiple-Dose Phase 1 Study to Evaluate the Safety and Pharmacokinetics of TAK-114 in Healthy Adult Japanese and Caucasian Male Subjects
Brief Title: TAK-114 Single- and Multiple-Dose Phase 1 Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-114/CPH-001; U1111-1162-6078 (Registry Identifier: WHO); JapicCTI-142691 (Registry Identifier: JapicCTI (Japan))
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Clinical Pharmacology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (15):
- Cohort 1A: TAK-114 10 mg (Experimental): Orally, once only.
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 1B: TAK-114 10 mg (Experimental): Orally, once
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 2A: TAK-114 20 mg (Experimental): Orally, once
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 2B: TAK-114 20 mg (Experimental): Orally, once
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 3A: TAK-114 50 mg (Experimental): Orally, once
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 3B: TAK-114 50 mg (Experimental): Orally, once
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 4a: TAK-114 20 mg (Experimental): Period 1: Single-dose administration in a fasting state Period 2: Single-dose administration 30 minutes after breakfast
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 4b: TAK-114 20 mg (Experimental): Period 1: Single-dose administration 30 minutes after breakfast Period 2: Single-dose administration in a fasting state
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 5A: TAK-114 20 mg (Experimental): Orally, Twice daily, 10 days
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 5B: TAK-114 20 mg (Experimental): Orally, Twice daily, 10 days
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 6A: TAK-114 50 mg (Experimental): Orally, Twice daily, 10 days
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 6B: TAK-114 50 mg (Experimental): Orally, Twice daily, 10 days
  Interventions: Drug: TAK-114 10 mg capsule
- Cohort 1A, 2A, 3A: TAK-114 placebo (Placebo Comparator): Cohort 1A, 2A, 3A: Orally, once
  Interventions: Drug: TAK-114 matched placebo
- Cohort 5A: TAK-114 placebo (Placebo Comparator): Cohort 5A: Orally, Twice daily, 10 days
  Interventions: Drug: TAK-114 matched placebo
- Cohort 6A: TAK-114 placebo (Placebo Comparator): Cohort 6A: Orally, Twice daily, 10 days
  Interventions: Drug: TAK-114 matched placebo

INTERVENTIONS:
Drug: TAK-114 10 mg capsule
  Arms: Cohort 1A: TAK-114 10 mg; Cohort 1B: TAK-114 10 mg; Cohort 2A: TAK-114 20 mg; Cohort 2B: TAK-114 20 mg; Cohort 3A: TAK-114 50 mg; Cohort 3B: TAK-114 50 mg; Cohort 4a: TAK-114 20 mg; Cohort 4b: TAK-114 20 mg; Cohort 5A: TAK-114 20 mg; Cohort 5B: TAK-114 20 mg; Cohort 6A: TAK-114 50 mg; Cohort 6B: TAK-114 50 mg
Drug: TAK-114 matched placebo
  Arms: Cohort 1A, 2A, 3A: TAK-114 placebo; Cohort 5A: TAK-114 placebo; Cohort 6A: TAK-114 placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of TAK-114 following single and multiple ascending oral doses in healthy Japanese male participants.

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blind, placebo-controlled, single and multiple oral dose study in healthy Caucasian and Japanese male participants.

The study is composed of three parts, Single-dose Ascending Part, Food Effect Part and Multiple-dose Ascending Part. Single-dose Ascending Part and Multiple-dose Ascending Part are designed as a randomized, double-blind or open-label, placebo-controlled, sequential-cohort, ascending single or multiple oral dose study of TAK-114 or matched placebo. The Food Effect Part is designed as a randomized, open-label, 2-period crossover study of a single dose of TAK-114.

ELIGIBILITY:
Inclusion Criteria:

Healthy Japanese participants:

* Must be willing to provide written informed consent and in the investigator's opinion able to comply with the study protocol.
* Is aged 20 to 45 years, inclusive.
* Weighs at least 50 kilogram (kg) and have a body mass index (BMI) between 18.5 and 25.0 kilogram per square meter (kg/m^2).

Healthy Caucasian participants:

* Must be willing to provide written informed consent and in the investigator's opinion able to comply with the study protocol.
* Is aged 20 to 45 years, inclusive; are of Caucasian descent (born to Caucasian parents and grandparents and has lived outside original country for less than 5 years) and maintains their original diet and lifestyle.
* Weighs at least 50 kg and have a body mass index between 18.5 and 30.0 kg/m2.

Exclusion Criteria:

• Participants have a known hypersensitivity to any component of the formulation of TAK-114 or any herb medicine or supplement related to Indigo naturalis.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Chair — Takeda
Locations (1):
- Sumida-ku, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 17 Nov 2014 to 29 April 2015.
Pre-assignment Details: Healthy Japanese, Caucasian participants enrolled in study with 3 parts to receive TAK-114 single rising dose (SRD) (10 milligram [mg], 20 mg and 50 mg, once daily) in Part 1, TAK-114 20 mg in fasted and fed conditions, cross-over in Period 1 and 2 of food effect Part 2 and TAK-114 multiple rising dose (MRD) (20 mg, 50 mg twice daily) in Part 3.
Groups:
- Part 1 SRD-Cohort 1A - 3A: Placebo: TAK-114 placebo-matching capsule, orally, once on Day 1 in the 3 days treatment period, in Japanese participants.
- Part 1 SRD-Cohort 1A: TAK-114 10 mg: TAK-114 10 mg, capsule, orally, once on Day 1 in the 3 days treatment period, in Japanese participants.
- Part 1 SRD-Cohort 2A: TAK-114 20 mg: TAK-114 20 mg, capsule, orally, once on Day 1 in the 3 days treatment period, in Japanese participants.
- Part 1 SRD-Cohort 3A: TAK-114 50 mg: TAK-114 50 mg, capsule, orally, once on Day 1 in the 3 days treatment period, in Japanese participants.
- Part 1 SRD - Cohort 1B : TAK-114 10 mg: TAK-114 10 mg, capsule, orally, once on Day 1 in the 3 days treatment period, in Caucasian participants.
- Part 1 SRD-Cohort 2B: TAK-114 20 mg: TAK-114 20 mg, capsule, orally, once on Day 1 in the 3 days treatment period, in Caucasian participants.
- Part 1 SRD-Cohort 3B: TAK-114 50 mg: TAK-114 50 mg, capsule, orally, once on Day 1 in the 3 days treatment period, in Caucasian participants.
- Part 2- Cohort 4: TAK-114 Fasted + TAK-114Fed: TAK-114 20 mg, capsule, orally, in fasted condition, once on Day 1 of Period 1 (3 days), followed by 14 days washout period, followed by TAK-114 20 mg, capsule, orally, in fed condition (after food), once on Day 1 of Period 2 (3 days), in Japanese participants.
- Part 2 Cohort 4: TAK-114 Fed + TAK-114 Fasted: TAK-114 20 mg, capsule, orally, in fed condition (after food), once on Day 1 of Period 2 (3 days), followed by 14 days washout period, followed by TAK-114 20 mg, capsule, orally, in fasted condition, once on Day 1 of Period 2 (3 days), in Japanese participants.
- Part 3 Placebo Cohort 5A - 6A: Placebo: TAK-114 placebo-matching, capsule, orally, twice daily on Days 1-9 and once only in the morning of Day 10 of the 10 days treatment period, in Japanese participants.
- Part 3 Cohort 5A MRD: TAK-114 20 mg: TAK-114 20 mg, capsule, orally, twice daily on Days 1-9 and once only in the morning of Day 10 of the 10 days treatment period, in Japanese participants.
- Part 3 Cohort 6A MRD: TAK-114 50 mg: TAK-114 50 mg, capsule, orally, twice daily on Days 1-9 and once only in the morning of Day 10 of the 10 days treatment period, in Japanese participants.
- Part 3 Cohort 5B MRD: TAK-114 20 mg: TAK-114 20 mg, capsule, orally, twice daily on Days 1-9 and once only in the morning of Day 10 of the 10 days treatment period, in Caucasian participants.
- Part 3 Cohort 6B MRD: TAK-114 50 mg: TAK-114 50 mg, capsule, orally, twice daily on Days 1-9 and once only in the morning of Day 10 of the 10 days treatment period, in Caucasian participants.
Period: All Parts (16 Days)
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2- Cohort 4: TAK-114 Fasted + TAK-114Fed | Part 2 Cohort 4: TAK-114 Fed + TAK-114 Fasted | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 6 | 6
Completed | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Only participants of Part 2 continued in next period.) | 6 (Only participants of Part 2 would continue in next period.) | 4 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).) | 6 (Participants from Part 1 and 3 did not continued in the washout period of Part 2 (crossover part).)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Crossover Period(Part 2:14 Days)
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2- Cohort 4: TAK-114 Fasted + TAK-114Fed | Part 2 Cohort 4: TAK-114 Fed + TAK-114 Fasted | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover Treatment (Part 2: 3 Days)
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2- Cohort 4: TAK-114 Fasted + TAK-114Fed | Part 2 Cohort 4: TAK-114 Fed + TAK-114 Fasted | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Groups:
- Part 2 Cohort 4: TAK-114 20 mg Fed + TAK-114 20 mg Fasted: TAK-114 20 mg, capsule, orally, once on Day 1, fed state in period 2 (3 days), followed by a 14 day washout period, further followed by TAK-114 20 mg, capsule, orally, once on Day 1 in fasted state in period 1, in healthy Japanese participants.
- Total: Total of all reporting groups
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2- Cohort 4: TAK-114 Fasted + TAK-114Fed | Part 2 Cohort 4: TAK-114 20 mg Fed + TAK-114 20 mg Fasted | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 31.5 (8.48) | 29.8 (7.25) | 28.3 (10.27) | 34.2 (10.26) | 32.0 (7.24) | 30.3 (5.65) | 26.3 (4.97) | 25.5 (3.51) | 35.3 (8.12) | 41.0 (4.08) | 30.3 (9.22) | 33.7 (10.73) | 29.3 (5.54) | 33.2 (5.74) | 31.3 (7.87)
Sex/Gender, Customized [Number; unit: Participants] — All participants enrolled in the study were male.
  Participants
    Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 82
Alcohol Classification [Number; unit: Participants]
  Drinks Every Day | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 7
  Drinks a Few Days per Week | 2 | 1 | 5 | 3 | 3 | 5 | 4 | 1 | 5 | 1 | 2 | 3 | 5 | 4 | 44
  Drinks a Few Days per Month | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 12
  Does not drink | 1 | 2 | 1 | 2 | 0 | 0 | 2 | 2 | 0 | 3 | 3 | 2 | 0 | 1 | 19
Caffeine Classification [Number; unit: Participants]
  Caffeine Consumption | 4 | 6 | 3 | 6 | 4 | 6 | 4 | 5 | 5 | 2 | 4 | 4 | 5 | 6 | 64
  No Caffeine Consumption | 2 | 0 | 3 | 0 | 2 | 0 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 0 | 18
Smoking Classification [Number; unit: Participants]
  Never smoked | 4 | 5 | 3 | 3 | 5 | 5 | 3 | 3 | 4 | 1 | 3 | 5 | 4 | 4 | 52
  Ex-smoker | 2 | 1 | 3 | 3 | 1 | 1 | 3 | 3 | 2 | 3 | 3 | 1 | 2 | 2 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE)
Time Frame: Baseline up to 3 days after the last dose of study drug (Day 3 in Part 1), (Day 20 in Part 2) and 7 days after the last dose of study drug (Day 17 in Part 3)
Population: The safety analysis set includes all participants who received the study drug.
Measure: Number; unit: participants
Groups:
- Part 2 Cohort 4: TAK-114 20 mg Fasted: TAK-114 20 mg, capsule, orally, in fasted condition, once on Day 1 of either Period 1 or 2 of 3 days, in Japanese participants.
- Part 2 Cohort 4: TAK-114 20 mg Fed: TAK-114 20 mg, capsule, orally, in fed condition (after food), once on Day 1 of either Period 1 or 2 of 3 days, in Japanese participants.
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2 Cohort 4: TAK-114 20 mg Fasted | Part 2 Cohort 4: TAK-114 20 mg Fed | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 12 | 4 | 6 | 6 | 6 | 6
participants | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 5 | 2 | 6

2. Primary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: Baseline up to Day 3 in Part 1, Day 20 in Part 2 and Day 17 in Part 3
Population: The safety analysis set includes all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2 Cohort 4: TAK-114 20 mg Fasted | Part 2 Cohort 4: TAK-114 20 mg Fed | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 12 | 4 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With TEAEs Related to Body Weight
Time Frame: Baseline up to Day 3 in Part 1, Day 20 in Part 2 and Day 17 in Part 3
Population: The safety analysis set includes all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2 Cohort 4: TAK-114 20 mg Fasted | Part 2 Cohort 4: TAK-114 20 mg Fed | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 12 | 4 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in 12-lead Electrocardiograms (ECG)
Description: Number of participants who had ECG shifts from "within normal limit" at baseline to "abnormal, clinically significant" after study drug administration were reported.
Time Frame: Baseline up to Day 3 in Part 1, Day 20 in Part 2 and Day 17 in Part 3
Population: The safety analysis set includes all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2 Cohort 4: TAK-114 20 mg Fasted | Part 2 Cohort 4: TAK-114 20 mg Fed | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 12 | 4 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in 12-lead Electrocardiograms (ECG)
Time Frame: Baseline up to Day 2 (only for Cohorts 1A, 2A, and 3A) in Part 1
Population: The safety analysis set includes all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants | 0 (0) | 0 (0) | 0 (0) | 0 (0)

6. Primary Outcome: Number of Participants With TEAEs Categorized Into Investigations System Organ Class (SOC) Related to Chemistry, Hematology or Urinalysis
Time Frame: Baseline up to Day 3 in Part 1, Day 20 in Part 2 and Day 17 in Part 3
Population: The safety analysis set includes all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2 Cohort 4: TAK-114 20 mg Fasted | Part 2 Cohort 4: TAK-114 20 mg Fed | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 12 | 4 | 6 | 6 | 6 | 6
participants
  C-reactive protein increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  White blood cell count increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood triglycerides increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Haemoglobin decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  High density lipoprotein decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

7. Secondary Outcome: Cmax - Maximum Observed Plasma Concentration for TAK-114
Time Frame: Day1: predose and at multiple time-points (up to 48 hours) postdose for Part 1; Day 1:predose and at multiple time-points (up to 48 hours) postdose in each period for Part 2; Day 10:predose and at multiple time points (up to 12 hours) postdose for Part 3
Population: The Pharmacokinetic (PK) analysis set includes all participants who had received the study drug and met the essential requirements defined in the study protocol without any critical protocol violations, and in whom PK assessment was possible.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2 Cohort 4: TAK-114 20 mg Fasted | Part 2 Cohort 4: TAK-114 20 mg Fed | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 12 | 6 | 5 | 6 | 3
picogram per milliliter (pg/mL) | 53.15 (10.051) | 68.74 (26.789) | 168.1 (71.210) | 30.98 (14.822) | 74.72 (17.886) | 140.8 (47.499) | 98.12 (34.944) | 150.8 (56.655) | 39.37 (4.8430) | 112.6 (12.857) | 24.53 (7.1949) | 106.7 (36.967)

8. Secondary Outcome: AUC (0-Infinity) - Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for Unchanged TAK-114: Part 1 and Part 2
Time Frame: Day 1: predose and at multiple time-points (up to 48 hours) postdose for Part 1; Day 1: predose and at multiple time-points (up to 48 hours) postdose in each period for Part 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: picogram*hour per milliliter (pg*hr/mL)
Arm/Group | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2 Cohort 4: TAK-114 20 mg Fasted | Part 2 Cohort 4: TAK-114 20 mg Fed
Number analyzed (Participants) | 6 | 5 | 6 | 3 | 5 | 6 | 12 | 12
picogram*hour per milliliter (pg*hr/mL) | 469.2 (112.44) | 762.2 (195.14) | 1708 (607.24) | 472.3 (77.694) | 879.2 (142.15) | 2180 (405.22) | 918.9 (165.75) | 918.2 (197.12)

9. Secondary Outcome: AUC (0-tau) - Area Under the Plasma Concentration-Time Curve From Time 0 to Time Tau for TAK-114: Part 3
Time Frame: Day10: predose and at multiple time points (up to 12 hours) postdose for Part 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 5 | 6 | 3
pg*hr/mL | 251.3 (47.209) | 838.0 (140.39) | 183.2 (49.061) | 749.7 (243.56)

10. Secondary Outcome: Mean Terminal Phase Elimination Half-life (T1/2) for TAK-114
Time Frame: Day1:predose and at multiple time-points (up to 48 hours) postdose for Part 1; Day1:predose and at multiple time-points (up to 48 hours) postdose in each period for Part 2; Day 10: predose and at multiple time points (up to 12 hours) postdose for Part 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2 Cohort 4: TAK-114 20 mg Fasted | Part 2 Cohort 4: TAK-114 20 mg Fed | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 5 | 6 | 3 | 5 | 6 | 12 | 12 | 6 | 5 | 6 | 3
hour | 4.108 (0.76763) | 5.500 (2.7925) | 5.272 (2.0918) | 7.417 (1.9012) | 5.822 (0.75503) | 6.213 (1.0856) | 4.294 (1.0600) | 3.705 (1.1044) | 4.972 (1.6574) | 6.970 (1.0813) | 6.045 (2.2456) | 7.283 (2.2407)

11. Secondary Outcome: Mean R(Cmax): Mean Accumulation Coefficient of Observed Maximum Plasma Concentration for TAK-114: Part 3
Description: Mean R(Cmax) was estimated as the ratio of Cmax on Day 10 and Cmax on Day 1. Cmax is the peak plasma drug concentration of TAK-114.
Time Frame: Days 1 and 10: predose and at multiple time points (up to 12 hours) postdose for Part 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 5 | 6 | 3
ratio | 0.2368 (0.05638) | 0.3606 (0.10037) | 0.2125 (0.06181) | 0.3190 (0.06630)

12. Secondary Outcome: Mean R(AUC): Mean of Accumulation Coefficient of Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-114: Part 3
Description: Mean R(AUC) was estimated as the ratio of AUC(0-tau) on Day 10 and AUC(0-tau) on Day 1. AUC (0-tau) is the area under the plasma concentration-time curve from time 0 to time tau.
Time Frame: Days 1 and 10: predose and at multiple time points (up to 12 hours) postdose for Part 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Number analyzed (Participants) | 6 | 5 | 6 | 3
ratio | 0.3032 (0.07024) | 0.4768 (0.15749) | 0.3128 (0.08596) | 0.4087 (0.04966)

13. Secondary Outcome: Urinary Excretion Ratio of TAK-114 From 0 to 48 Hours Postdose: Part 1
Description: Urinary excretion ratio (% of dose) of TAK-114 in urine were calculated for each participant. Ratio was calculated from the urine concentrations of each analyte and the volume of urine collected.
Time Frame: Day 1: 0 to 48 hours postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6
percentage of dose | 0.003835 (0.0019990) | 0.001984 (0.00055667) | 0.002759 (0.0017349) | 0.003724 (0.0022022) | 0.003143 (0.00083500) | 0.002420 (0.0012154)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after first dose of study drug and no more 3 days after the last dose of study drug (Day 3 in Part 1), (Day 20 in Part 2) and 7 days after the last dose of study drug (Day 17 in Part 3).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1 SRD-Cohort 1A - 3A: Placebo | Part 1 SRD-Cohort 1A: TAK-114 10 mg | Part 1 SRD-Cohort 2A: TAK-114 20 mg | Part 1 SRD-Cohort 3A: TAK-114 50 mg | Part 1 SRD - Cohort 1B : TAK-114 10 mg | Part 1 SRD-Cohort 2B: TAK-114 20 mg | Part 1 SRD-Cohort 3B: TAK-114 50 mg | Part 2 Cohort 4: TAK-114 20 mg Fasted | Part 2 Cohort 4: TAK-114 20 mg Fed | Part 3 Placebo Cohort 5A - 6A: Placebo | Part 3 Cohort 5A MRD: TAK-114 20 mg | Part 3 Cohort 6A MRD: TAK-114 50 mg | Part 3 Cohort 5B MRD: TAK-114 20 mg | Part 3 Cohort 6B MRD: TAK-114 50 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/12 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 1/6 | 1/6 | 0/6 | 1/6 | 0/12 | 1/12 | 0/4 | 3/6 | 5/6 | 2/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 SRD-Cohort 1A - 3A: Placebo (N=6) | Part 1 SRD-Cohort 1A: TAK-114 10 mg (N=6) | Part 1 SRD-Cohort 2A: TAK-114 20 mg (N=6) | Part 1 SRD-Cohort 3A: TAK-114 50 mg (N=6) | Part 1 SRD - Cohort 1B : TAK-114 10 mg (N=6) | Part 1 SRD-Cohort 2B: TAK-114 20 mg (N=6) | Part 1 SRD-Cohort 3B: TAK-114 50 mg (N=6) | Part 2 Cohort 4: TAK-114 20 mg Fasted (N=12) | Part 2 Cohort 4: TAK-114 20 mg Fed (N=12) | Part 3 Placebo Cohort 5A - 6A: Placebo (N=4) | Part 3 Cohort 5A MRD: TAK-114 20 mg (N=6) | Part 3 Cohort 6A MRD: TAK-114 50 mg (N=6) | Part 3 Cohort 5B MRD: TAK-114 20 mg (N=6) | Part 3 Cohort 6B MRD: TAK-114 50 mg (N=6)
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
High density lipoprotein decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.